CLINICAL TRIAL: NCT04770740
Title: A Phase 2, Double Blind, Randomized, Placebo-controlled Clinical Trial to Investigate the Safety and Effects of Oral Vitamin K2 Supplementation in COVID-19
Brief Title: Randomized Controlled Clinical Trial to Investigate Effects of Vitamin K2 in COVID-19
Acronym: KOVIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Canisius-Wilhelmina Hospital (Other)
Collaborators: Kappa Bioscience AS (Unknown)
Responsible Party: Principal Investigator, Ton Dofferhoff, Specialist in Internal Medicine and infectious diseases, Canisius-Wilhelmina Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: KOVIT
Record Dates: First submitted 2021-02-24; First posted 2021-02-25 (Actual); Last update posted 2022-06-13 (Actual); Status verified 2022-06

CONDITIONS: Covid19
Keywords: Vitamin K; Desmosine; Elastic fibers; Dp-ucMGP; PIVKA-II
MeSH Terms: conditions — COVID-19 | interventions — Vitamin K 2

STUDY DESIGN:
Intervention Model Description: double blind, randomized, placebo-controlled (phase 2)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Vitamin K2 (Active Comparator): Patients with COVID-19 who get our dietary supplement vitamin K2, three tablets of 333mcg a day, for 14 days or until discharge, whichever occurs earlier.
  Interventions: Dietary Supplement: Vitamin K2 in the form of Menaquinone-7 (MK-7)
- Control: Placebo (Placebo Comparator): Patients with COVID-19 who get placebo as control, three tablets a day, for 14 days or until discharge, whichever occurs earlier.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vitamin K2 in the form of Menaquinone-7 (MK-7) — Patients will take three tablets of vitamin K2 menaquinone-7 (333mcg) per day. Patients taking vitamin K2 MK-7 will receive the total of 999mcg per day from day 1 until day 14 or discharge, whichever occurs earlier. All subjects can be treated with prophylactic or therapeutic heparin-based (heparin or any low-molecular weight heparin) anticoagulants, according to local hospital protocols. Provided by Kappa Bioscience.
  Arms: Experimental: Vitamin K2
Dietary Supplement: Placebo — Patients will take three tablets of placebo containing only inactive ingredients per day, from day 1 until day 14 or until discharge, whichever occurs first. The placebo is provided by Kappa Bioscience.
  Arms: Control: Placebo

SUMMARY:
Coronavirus disease 2019 (COVID-19) is caused by the severe acute respiratory syndrome coronavirus-2 (SARS-CoV-2). While the majority of people recover after mild symptoms, a portion of COVID-19 patients develops respiratory failure. Coagulopathy and thromboembolism are prevalent in severe COVID-19, and these factors are associated with decreased survival. Coagulation is an intricate balance between clot promoting and dissolving processes in which vitamin K plays an essential role. Elastin is a major component of dynamic tissues such as lungs and arteries, and elastin calcification stimulates elastin degradation and vice versa. The vitamin K-dependent Matrix Gla Protein (MGP) protects elastin from both calcification and degradation.

Although technically feasible, direct quantification of blood vitamin K levels is not an appropriate method to assess overall vitamin K status due to differences in bioavailability and half-life time between the two naturally occurring vitamin K forms (vitamin K1 and K2). Measuring inactive levels of vitamin K-dependent proteins in the circulation is the method recommended by most experts, as it represents the systemic availability of both vitamin K1 and K2. Dp-uc (dephospho uncarboxylated, i.e. inactive) MGP and proteins induced by vitamin K absence (PIVKA-II) both inversely correlate with vitamin K status and can be used as surrogate markers of total vitamin K status.

Recently, we found a severely reduced vitamin K status (as quantified by dp-ucMGP) in COVID-19 patients compared to controls. In COVID-19 patients, low vitamin K status was also associated with poor outcome (defined as the need for invasive ventilation or death), accelerated elastin degradation (quantified by plasma (iso)desmosine (DES) a byproduct of elastin degradation). Based on these finding and previous studies, we hypothesize that improving vitamin K-status by vitamin K supplementation could have favorable effects on pulmonary damage and coagulopathy in COVID-19.

DETAILED DESCRIPTION:
The outbreak of coronavirus 2019 disease (COVID-19) has a major impact on health care worldwide. This infectious disease is caused by the severe acute respiratory syndrome coronavirus (SARS-CoV-2). The majority of individuals who contract COVID-19 have mild symptoms, but a significant part develops respiratory failure due to severe pneumonia and/or acute respiratory distress syndrome (ARDS). The virus may also have extra pulmonary manifestations, including coagulopathy and venous thromboembolism, associated with decreased survival. The pathogenesis of this coagulopathy, and the links between pulmonary and thromboembolic manifestations of COVID-19 are incompletely understood. In KOVIT trial, the roll of vitamin K in the pathogenesis of these manifestations will be elucidated.

Vitamin K in coagulation and elastic fiber metabolism

Coagulation is an intricate balance between clot promoting and dissolving processes in which vitamin K plays an important role. Pro-coagulation factors II, VII, IX and X depend on vitamin K for carboxylation to fulfill their biological function. Besides this, vitamin K is also cofactor of anticoagulant protein C and protein S. A significant proportion of protein S is extrahepatically synthesized in endothelial cells, in contrast to the pro-coagulant factors and protein C. Protein S plays a local suppressive role against thrombosis.

Matrix Gla protein (MGP) is also vitamin K-dependent but not involved in intravascular coagulation. MGP has been generally studied as an inhibitor of vascular mineralization, and its role in the pulmonary compartment seems to be comparable. Besides preventing soft tissue calcification, it also protects against elastic fiber degradation. Elastic fibers are fundamental matrix components in lungs and have high calcium affinity. Degradation and mineralization of elastic fibers are related processes. Desphospho-uncarboxylated MGP (dp-ucMGP) i.e. inactive MGP is a robust biomarker of extrahepatic vitamin K status since it is inversely associated with vitamin K.

Insufficiency of vitamin K may develop within days of poor intake, particularly in pathological conditions of increased vitamin K utilization. During times of scarcity, micronutrients are reserved for use in processes that form the greatest threat to short-term survival. With regard to vitamin K insufficiency, it appears to be preferentially transported to the liver for the activation (via carboxylation) of procoagulant factors at the expense of extrahepatic vitamin K-dependent proteins such as MGP and protein S (figure 1).

Assessment of vitamin K status

In nature, vitamin K is found in food as vitamin K1 (phylloquinone) and vitamin K2 (menaquinones). Measuring circulating levels of these two forms of vitamin K is technically feasible but the value of such measurements is limited. Quantification of vitamin K-dependent proteins that have not been carboxylated yet, is a valuable method reflecting the functional deficit of vitamin K1 and K2. Determination of dp-ucMGP levels as well as the ratio between uncarboxylated and carboxylated osteocalcin are validated assays of extrahepatic vitamin K status.

Dp-ucMGP is a biomarker of extrahepatic vitamin K status. High dp-ucMGP reflects low vitamin K status and vice versa. Although increasing vitamin K consumption decreases the amount of dp-ucMGP. Circulating dp-ucMGP concentration can best be regarded as a reflection of the total extrahepatic vitamin K deficit, which refers to the amount of vitamin K that is needed to carboxylate all the uncarboxylated vitamin K-dependent proteins in the body. Hepatic vitamin K status is usually quantified by measuring levels of protein induced by vitamin K absence (PIVKA)-II (i.e. uncarboxylated prothrombin).

Rationale for study treatment

Recently, a reduced vitamin K status was found, as quantified by dp-ucMGP, in patients suffering from COVID-19 as compared to controls. In these patients, low vitamin K status was also associated with poor outcome (defined as the need for invasive ventilation or death) and accelerated elastic fiber degradation (quantified by plasma (iso)desmosine (DES) a byproduct of elastin degradation). In contrast, hepatic vitamin K status, measured by inactive factor II (also called protein-induced by vitamin K absence (PIVKA)-II) was unaffected in most patients (figure 2). Considering the preferential activation of hepatic over extrahepatic proteins.

In COVID-19, inflammation causes pulmonary elastic fiber damage, which could also lead to an upregulation of MGP and a draining of extrahepatic vitamin K. The significant correlation between increased dp-ucMGP levels, and elastic fiber degeneration and poor prognosis supports the theory that vitamin K insufficiency contributes to pulmonary pathology.

Hypothesis

It is hypothesized that improving vitamin K-status by vitamin K supplementation could have favorable effects on both pulmonary damage and coagulation abnormalities in COVID-19 patients.

Objective

The objective of the KOVIT trial is to evaluate the safety of oral vitamin K2 supplementation in patients suffering from COVID-19 requiring hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* COVID-19 patients who are admitted to the CWZ with COVID-19, with a laboratory confirmed SARS-CoV-2 infection within the previous 96 hours
* Respiratory failure requiring supplemental oxygen, defined as requiring supplemental oxygen to sustain an arterial PO2 ≥70mmHg (measured by arterial blood gas) or an oxygen saturation of ≥94% (measured using a pulse oximeter)
* At least 18 years old
* Able to safely swallow the study medication or possibility of safely administering this through a nasogastric tube
* Use of prophylactic heparin or LWMH according to hospital protocols, or use of therapeutic dosages if there is a medical indication for this
* Informed consent signed by patient

Exclusion Criteria:

* Use of oral anticoagulation drugs; patients may be included when they have been switched to LMWH
* Patients on vitamin K antagonists with a supra-therapeutic anticoagulation at admission who require vitamin K supplementation to correct this, or were administered vitamin K for this reason within the preceding 5 days
* Patients already using vitamin K supplements at admission
* Participation in another intervention study
* Direct admission to an intensive care unit (ICU) for invasive ventilation at presentation
* Confirmed active pulmonary embolism or deep venous thrombosis prior to inclusion
* Known allergy to any of the components of the study medication or placebo
* Patients who are hemodialysis dependent at admission
* Pregnancy at the time of inclusion
* Diagnosed malignancy at the time of inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-03-01 (Actual)

PRIMARY OUTCOMES:
Plasma desmosine levels | Day 1 until day 28 or until discharge if this is earlier.
  Plasma desmosine levels before and during vitamin K supplementation in intervention versus control patients.
Plasma dp-ucMGP levels | Day 1 until day 28 or until discharge if this is earlier.
  Plasma dp-uc MGP levels before and during vitamin K supplementation within the intervention group and in intervention versus control patients.

SECONDARY OUTCOMES:
Difference between the number of grade 3 and grade 4 adverse events | Day 1 until day 28
  Difference between the number of grade 3 and grade 4 adverse events between the intervention and control group during treatment, with special attention for: progression of respiratory insufficiency, thrombotic events, pulmonary embolism or deep venous thrombosis, bleeding, renal insufficiency, cardiac decompensation, liver enzyme abdnormalities and/or liver failure.
Serum PIVKA-II levels | Day 1 until day 28 or until discharge if this is earlier.
  Serum PIVKA-II levels before and during vitamin K supplementation in intervention versus control patients.

CONTACTS AND LOCATIONS:
Overall Officials: A. Dofferhoff, M.D. PhD, Principal Investigator — Canisius-Wilhelmina Hospital
Locations (1):
- Canisius Wilhelmina Hospital, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
Not sure yet.

REFERENCES:
- [Background] Janssen R, Visser MPJ, Dofferhoff ASM, Vermeer C, Janssens W, Walk J. Vitamin K metabolism as the potential missing link between lung damage and thromboembolism in Coronavirus disease 2019. Br J Nutr. 2021 Jul 28;126(2):191-198. doi: 10.1017/S0007114520003979. Epub 2020 Oct 7. PMID 33023681
- [Background] Dofferhoff ASM, Piscaer I, Schurgers LJ, Visser MPJ, van den Ouweland JMW, de Jong PA, Gosens R, Hackeng TM, van Daal H, Lux P, Maassen C, Karssemeijer EGA, Vermeer C, Wouters EFM, Kistemaker LEM, Walk J, Janssen R. Reduced Vitamin K Status as a Potentially Modifiable Risk Factor of Severe Coronavirus Disease 2019. Clin Infect Dis. 2021 Dec 6;73(11):e4039-e4046. doi: 10.1093/cid/ciaa1258. PMID 32852539
- See also: Kappa Bioscience — https://www.kappabio.com/